CLINICAL TRIAL: NCT04726371
Title: Best Practices to Prevent COVID-19 Illness in Staff and People With Serious Mental Illness and Developmental Disabilities in Congregate Living Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Advocates (Unknown); Bay Cove Human Services (Other); North Suffolk Mental Health Association (Other); Open Sky Community Services (Unknown); Riverside Community Care, Inc. (Unknown); Dartmouth College (Other); Vinfen (Industry)
Responsible Party: Principal Investigator, Stephen Bartels, Director, The Mongan Institute; James J. and Jean H. Mongan Chair of Health Policy and Community Health; Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P003803, 2020P003957
Record Dates: First submitted 2021-01-15; First posted 2021-01-27 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Intellectual Disability; Developmental Disability; Axis I Diagnosis; Mental Illness; Covid19; Coronavirus
Keywords: COVID-19; Coronavirus; Intellectual Disabilities; Developmental Disabilities; Serious Mental Illness; Congregate Living; Group Homes
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities; Mental Disorders; COVID-19; Coronavirus Infections | interventions — tributyl phosphate

STUDY DESIGN:
Intervention Model Description: The investigators will employ a cluster-randomized trial design with ~200 group homes randomized to the implementation of "Tailored Best Practices" (TBP) compared to ~200 group homes randomized to "Generic Best Practices" (GBP). Randomization will occur at the level of the group home stratified by group home type (SMI versus ID/DD), incident COVID-19 infection in the staff and residents (high incidence versus low incidence), and race/ethnicity (proportion non-Hispanic Caucasian versus other). TBP and GBP will be delivered within each agency as part of routine training activities. TBP sites will receive coaching specific to the setting, staff, and residents. The best practice implementation fidelity (i.e. staff and residents participating in recommended screening, isolating, contact tracing, PPP protocols, and vaccine acceptance), and COVID-19 incidence are co-primary outcomes with group home as the unit of analysis. The outcomes will be assessed at baseline, 3, 6, 9, 12, and 15 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generic Best Practices (GBP) (Active Comparator): The ~200 group homes randomized into this arm will receive the Generic Best Practices (GBP) intervention package as part of routine training activities. GBP consists of state and federal standard guidelines for COVID-19 mitigation for all congregate living settings.
  Interventions: Behavioral: Generic Best Practices
- Tailored Best Practices (TBP) (Experimental): The ~200 group homes randomized into this arm will receive the Tailored Best Practices (TBP) intervention package as part of routine training activities. TBP consists of COVID-19 mitigation measures specifically adapted for staff and residents with SMI and ID/DD in congregate living settings. Sites in this arm will receive coaching specific to the setting, staff, and residents.
  Interventions: Behavioral: Tailored Best Practices

INTERVENTIONS:
Behavioral: Generic Best Practices — GBP consists of (1) Massachusetts Executive Office of Health and Human Services distribution of standard guidelines and policies for public health prevention and management of COVID and (2) standard virtual training of the staff of the group homes in these generic COVID-19 prevention practices including recommended use of hand washing, use of PPE, and symptom-triggered screening. Group homes randomized to this intervention will receive standard recommended and fully vetted best practices with respect to preventing and managing COVID-19 based on recommendations by the CDC and on consultation with leading national experts in infectious disease working with the Commonwealth of Massachusetts. The control condition does not represent inferior or substandard practice. As findings occur and as policy leads to adjustments in recommendations during the course of the study, the GBP condition will incorporate recommendations that are appropriate and up-to-date with CDC and state policy.
  Other Names: GBP
  Arms: Generic Best Practices (GBP)
Behavioral: Tailored Best Practices — TBP consists of optimized, tailored, and highly specific COVID-19 best practices and training materials specific to the setting, staff, and residents with SMI and ID/DD in congregate living settings based on the comparative effectiveness of different types, intensities, and combinations of COVID-19 prevention practices (screening, isolation, contact tracing, use of PPP, vaccination) specifically modeled for residents and staff of congregate living settings for people with ID/DD and SMI derived by a simulation model. Results from this modeling process will be provided to stakeholders to support decision makers in prioritizing resources and practices with the greatest impact on reducing COVID-19 tailored for people with SMI and ID/DD in congregate living settings. This process to determine the content of TBP will occur as part of this study prior to randomization.
  Other Names: TBP
  Arms: Tailored Best Practices (TBP)

SUMMARY:
Best Practices to Prevent COVID-19 Illness in Staff and People With Serious Mental Illness and Developmental Disabilities in Congregate Living Settings is a research study aimed at developing, implementing, and evaluating a package of interventions specifically designed to reduce COVID-19 and other infectious-disease incidence, hospitalizations, and mortality among staff and adults with Serious Mental Illness and Intellectual and Developmental Disabilities in congregate-living settings.

DETAILED DESCRIPTION:
Persons with Serious Mental Illness (SMI) and Intellectual Disabilities and Developmental Disabilities (ID/DD) are disproportionately vulnerable to COVID-19 for three reasons: (1) Medical vulnerability. Smoking, chronic obstructive pulmonary disease, cardiovascular disease, and diabetes all increase COVID-19 mortality and are about 2-3 times more prevalent among persons with SMI. People with ID/DD suffer higher rates of COVID-19 risk factors, including pre-existing chronic conditions, heart defects, obesity, chronic respiratory problems or lung disease, lower immune function, cancer, and diabetes. (2) Residential vulnerability. The congregate care settings in which many people with SMI and ID/DD live carry many of the same higher risks of COVID-19 transmission currently affecting assisted-living settings and nursing homes across the nation. (3) Health behavior vulnerability. Some people with SMI and ID/DD have cognitive, behavioral, and physical challenges that heighten COVID-19 risk by hampering personal protective practices (PPP) (i.e., hand hygiene, physical distancing, use of face masks). Moreover, the staff who work in congregate care settings are often subject to high rates of exposure, have low socioeconomic status, use public transportation, and lack personal protective equipment. This collection of factors contributes to an extraordinarily high risk of COVID-19 morbidity, and mortality. Despite payment reforms and mandated best practices for COVID-19 for congregate care by the MA Department of Public Health, rates of coronavirus illness for residents with SMI and ID/DD are 8 times higher (12%), and for staff 2 times higher (3.0%), compared to the general population in the surrounding "hot spot" communities (1.5%) selected for this study. This tragic health disparity confirms that key decision-makers lack the knowledge of how to optimally tailor best practices for this highly vulnerable population and the staff who provide their care to effectively reduce their high risk of COVID-19 and COVID-19 related mortality.

The investigators' overall goal is to reduce COVID-19 and other infectious-disease incidence, hospitalizations, and mortality among staff and adults with Serious Mental Illness (SMI) and Intellectual and Developmental Disabilities (ID/DD) in congregate-living settings in Massachusetts. The investigators address 2 comparative-effectiveness questions:

With the goal of prioritizing and resourcing actionable best practices: What is the comparative effectiveness of different types and intensities of five basic preventive interventions-screening, isolation, contact tracing, personal protective practices (PPP) (i.e., hand hygiene, physical distancing, use of face masks), and vaccination-in reducing rates of COVID-19, hospitalizations, and mortality in staff and adult residents with SMI and ID/DD in congregate care settings? Effectiveness Hypothesis: Of the 5 preventive interventions, tailored screening, effective use of isolation, and increased vaccination acceptance will be associated with the greatest reduction of staff and resident COVID-19 rates and related hospitalizations.

With the goal of effectively implementing best practices: What is the most effective implementation strategy to reduce rates of COVID-19 in congregate care settings for persons with SMI and ID/DD: (1) Tailored Best Practices (TBP) specifically adapted for staff and residents with SMI and ID/DD in congregate living settings or (2) Generic Best-Practices (GBP) consisting of state and federal standard guidelines for all congregate care settings? Implementation Hypothesis: TBP will be associated with greater implementation fidelity and lower staff and resident rates of COVID-19 and hospitalization than GBP.

To test these hypotheses, the investigators will pursue three Aims:

Aim 1: The investigators will synthesize existing data collected by the six provider organizations on (1) rates of COVID-19, hospitalization, and mortality and (2) use of screening, isolation, contact tracing, PPP, and vaccination in 400 group homes for SMI and ID/DD. The investigators will also collect qualitative data through surveys and virtual focus groups on the experience of staff and residents, and on barriers and facilitators to implementing recommended practices.

Aim 2: The investigators will determine the comparative effectiveness of different COVID-19 preventive practices (screening, isolation, contact tracing, use of PPP, vaccination) by populating a validated simulation model and engage decision makers and stakeholders in selecting priorities for best practices. The investigators will apply the Clinical and Economic Analysis of COVID-19 Interventions (CEACOV), a COVID-19 simulation model that has already been developed and validated, to simulate the 2,050 residents and 3,300 staff of the 400 group homes for persons with SMI and ID/DD in the study. The investigators will compare the effectiveness of different types, intensities, and combinations of the five identified interventions: screening, isolation, contact tracing, PPP, and vaccination.

On completion of the simulation modeling at month 3, the investigators will convene a COVID-19 Quality Improvement Collaborative (CQIC) Virtual Summit including consumers, providers, advocates, and key decision makers, during which the investigators will summarize the results of the comparative effectiveness simulation model and present alternative scenarios demonstrating the impact of increasing or decreasing amounts or combinations of various practices. The CQIC Virtual Summit and 1-2 additional brief virtual meetings will result in recommendations for a final prioritized set of actionable and feasible Tailored Best Practices (TBP) for implementation. The CQIC will review and adapt relevant COVID-19 training materials and finalize a TBP implementation package.

Aim 3: The investigators will employ a cluster randomized trial design with 200 group homes randomized to implementation of "Tailored Best Practices" (TBP) compared to 200 group homes randomized to "Generic Best Practices" (GBP). The investigators will engage in a three-month observational pre-randomization period to assess the baseline use of preventive practices and rates of COVID in each group home to better isolate the effect of the introduction of the TBP intervention. The investigators have also incorporated a 3-month implementation phase in order to accommodate implementing the TBP intervention with fidelity across 200 group homes during the same time period. The best practice implementation fidelity and COVID-19 incidence are co-primary outcomes with group home as the unit of analysis. Within each site, the investigators will engage in repeated measurement of these outcomes across 6 time points (Baseline, 3, 6, 9, 12, and 15 months) so that time effects (observed and latent) can be modeled precisely in the presence of any fluctuations in incidence over time.

By month 16 of the project, the investigators will know the effectiveness of the Tailored Best Practices (TBP) implementation for a diverse array of state-supported group homes for SMI and ID/DD with broad generalizability to similar settings across the nation that will be broadly distributed through dissemination materials at the end of the project.

ELIGIBILITY:
Inclusion Criteria:

1. All congregate care homes in Massachusetts operated by the following public-sector community-based human service organizations: Vinfen, Bay Cove, Advocates, North Suffolk, Open Sky, and Riverside
2. The group home must serve adults with SMI (Serious Mental Illness, i.e., DSM-V Diagnosis of Axis-I Mental Illness with persistent functional impairment) or adults with ID/DD (Intellectual and Developmental Disabilities)
3. All residents and staff of the home must be age 18 or older

Exclusion Criteria:

1. All congregate care homes in Massachusetts not operated by any of the public-sector community-based human service organizations mentioned above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bartels, MD, MS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bartels S, Levison JH, Trieu HD, Wilson A, Krane D, Cheng D, Xie H, Donelan K, Bird B, Shellenberger K, Cella E, Oreskovic NM, Irwin K, Aschbrenner K, Fathi A, Gamse S, Holland S, Wolfe J, Chau C, Adejinmi A, Langlois J, Reichman JL, Iezzoni LI, Skotko BG. Tailored vs. General COVID-19 prevention for adults with mental disabilities residing in group homes: a randomized controlled effectiveness-implementation trial. BMC Public Health. 2024 Jun 26;24(1):1705. doi: 10.1186/s12889-024-18835-w. PMID 38926810
- [Derived] Becker JE, Shebl FM, Losina E, Wilson A, Levison JH, Donelan K, Fung V, Trieu H, Panella C, Qian Y, Kazemian P, Bird B, Skotko BG, Bartels S, Freedberg KA. Using simulation modeling to inform intervention and implementation selection in a rapid stakeholder-engaged hybrid effectiveness-implementation randomized trial. Implement Sci Commun. 2024 Jun 24;5(1):70. doi: 10.1186/s43058-024-00593-w. PMID 38915130
- [Derived] Constantin AM, Noertjojo K, Sommer I, Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, McElvenny DM, Rhodes S, Martin C, Sampson O, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD015112. doi: 10.1002/14651858.CD015112.pub3. PMID 38597249
- [Derived] Fung V, Levison JH, Wilson A, Cheng D, Chau C, Krane D, Trieu HD, Irwin K, Cella E, Bird B, Shellenberger K, Silverman P, Batson J, Fathi A, Gamse S, Wolfe J, Holland S, Donelan K, Samuels R, Becker JE, Freedberg KA, Reichman JL, Keller T, Tsai AC, Hsu J, Skotko BG, Bartels S. COVID-19-Related Outcomes Among Group Home Residents with Serious Mental Illness in Massachusetts in the First Year of the Pandemic. Adm Policy Ment Health. 2024 Jan;51(1):60-68. doi: 10.1007/s10488-023-01311-9. Epub 2023 Nov 8. PMID 37938475
- [Derived] Levison JH, Krane D, Donelan K, Aschbrenner K, Trieu HD, Chau C, Wilson A, Oreskovic NM, Irwin K, Iezzoni LI, Xie H, Samuels R, Silverman P, Batson J, Fathi A, Gamse S, Holland S, Wolfe J, Shellenberger K, Cella E, Bird B, Skotko BG, Bartels S. Best practices to reduce COVID-19 in group homes for individuals with serious mental illness and intellectual and developmental disabilities: Protocol for a hybrid type 1 effectiveness-implementation cluster randomized trial. Contemp Clin Trials. 2023 Feb;125:107053. doi: 10.1016/j.cct.2022.107053. Epub 2022 Dec 17. PMID 36539061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Unit of recruitment and analysis was Group Home (GH). Recruitment occurred between 11/2020-12/2020. CEOs of 6 provider organizations provided letters of commitment to participate in the trial and written consent for their sites to be included. All GHs were included other than those with residents <=18 years of age and Acquired Brain Injury homes. No individual participants were recruited, provided informed consent, or were enrolled in the study.
Pre-assignment Details: No group homes enrolled in the study were excluded before assignment to groups.
Units Other Than Participants: Group home
Groups:
- Generic Best Practices (GBP): The 207 group homes randomized into this arm received the Generic Best Practices (GBP) intervention package as part of routine training activities. GBP consisted of state and federal standard guidelines for COVID-19 mitigation for all congregate living settings.
  Generic Best Practices: GBP consisted of (1) Massachusetts Executive Office of Health and Human Services distribution of standard guidelines and policies for public health prevention and management of COVID and (2) standard virtual training of the staff of the group homes in these generic COVID-19 prevention practices including recommended use of hand washing, use of PPE, and symptom-triggered screening. Group homes randomized to this intervention received standard recommended and fully vetted best practices with respect to preventing and managing COVID-19 based on recommendations by the CDC and on consultation with leading national experts in infectious disease working with the Commonwealth of Massachusetts. The control condition did not represent inferior or substandard practice. As findings occurred and as policy led to adjustments in recommendations during the course of the study, the GBP condition incorporated recommendations that were appropriate and up-to-date with CDC and state policy.
- Tailored Best Practices (TBP): The 208 group homes randomized into this arm received the Tailored Best Practices (TBP) intervention package as part of routine training activities. TBP consisted of COVID-19 mitigation measures specifically adapted for staff and residents with SMI and ID/DD in congregate living settings. Sites in this arm received coaching specific to the setting, staff, and residents.
  Tailored Best Practices: TBP consisted of optimized, tailored, and highly specific COVID-19 best practices and training materials specific to the setting, staff, and residents with SMI and ID/DD in congregate living settings based on the comparative effectiveness of different types, intensities, and combinations of COVID-19 prevention practices (screening, isolation, contact tracing, use of PPP, vaccination) specifically modeled for residents and staff of congregate living settings for people with ID/DD and SMI derived by a simulation model. There were four main components to Tailored Best Practices: Measurement, Feedback, and House Plans; Motivational Interviewing; Interactive Education; and Trusted Messengers.
Period: Overall Study
Arm/Group | Generic Best Practices (GBP) | Tailored Best Practices (TBP)
Started | 4836; 207 Group home | 4538; 208 Group home
Residents (Vaccination Analysis) (The sample used for vaccination analysis was limited to individuals who were not fully vaccinated at baseline. This is a subsample of the sample used for the COVID-19 incidence and fidelity primary analyses.) | 492; 207 Group home | 407; 208 Group home
Staff (Vaccination Analysis) (The sample used for vaccination analysis was limited to individuals who were not fully vaccinated at baseline. This is a subsample of the sample used for the COVID-19 incidence and fidelity primary analyses.) | 836; 207 Group home | 836; 208 Group home
Completed | 3481; 206 Group home | 3262; 208 Group home
Not Completed | 1355; 1 Group home | 1276; 0 Group home

BASELINE CHARACTERISTICS:
Population: Due to our project design, 2,345 participants had delayed entry to the study. As the unit of randomization was the group home and not individual participants, this was a dynamic sample. The Participant Flow reflects all participants who entered the study at any point. The Baseline Analysis Population reflects only those participants present during the baseline period of the study.
Units Other Than Participants: Group homes
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Best Practices (GBP) | Tailored Best Practices (TBP) | Total
Number analyzed (Participants) | 3,600 | 3,429 | 7,029
Number analyzed (Group homes) | 207 | 208 | 415
Age, Continuous [Mean (Standard Deviation); unit: years]
  number analyzed (Participants) | 3,600 | 3,429 | 7029
  (all) | 44.54 (5.90) | 44.16 (5.84) | 44.36 (5.87)
Sex/Gender, Customized [Mean (Standard Deviation); unit: percentage of participants]
  number analyzed (Participants) | 3,600 | 3,429 | 7029
  Female | 48.74 (23.48) | 49.53 (23.86) | 49.13 (23.65)
  Male | 49.87 (23.45) | 49.20 (23.78) | 49.54 (23.59)
  Other/missing | 1.40 (3.75) | 1.27 (3.28) | 1.33 (3.52)
Race/Ethnicity, Customized [Mean (Standard Deviation); unit: percentage of participants]
  number analyzed (Participants) | 3,600 | 3,429 | 7029
  NH White | 38.39 (22.45) | 35.70 (22.21) | 37.06 (22.35)
  NH Black or African-American | 48.01 (22.72) | 51.08 (22.94) | 49.53 (22.86)
  Hispanic/Latinx | 4.70 (6.41) | 5.06 (7.72) | 4.88 (7.08)
  NH Other | 4.16 (6.90) | 4.37 (7.27) | 4.26 (7.08)
  Not answered/Missing | 4.73 (7.12) | 3.79 (6.16) | 4.26 (6.67)
Division [Count of Units; unit: Group homes]
  number analyzed (Participants) | 3,600 | 3,429 | 7029
  ID/DD | 103 | 103 | 206
  SMI | 104 | 105 | 209

OUTCOME MEASURES:

1. Primary Outcome: New COVID-19 Group Home Incidence
Description: New laboratory-confirmed COVID-19 cases among residents and staff. Measured as new cases per 100 person-months.
Time Frame: The outcome was measured at baseline, 3-, 6-, 9-, 12-, and 15-months post-baseline.
Population: One group home in the GBP arm closed between the 6- and 9-month follow-up periods. The BL sample size here is different than the BL descriptive table. For the BL descriptive table, we assigned participants on an intent-to-treat basis in order to avoid overlap. However, for our analysis, participant allocation was based on the home that they lived or worked in during the study period. Since some staff worked in multiple homes across both arms, the samples are not mutually exclusive.
Measure: Mean (95% Confidence Interval); unit: New COVID-19 cases per 100 person-months
Units Other Than Participants: Group home
Arm/Group | Generic Best Practices (GBP) | Tailored Best Practices (TBP)
Number analyzed (Participants) | 4,867 | 4,507
Number analyzed (Group home) | 207 | 208
New COVID-19 cases per 100 person-months
  Baseline: number analyzed (Participants) | 3960 | 3756
  Baseline | 1.61 [1.38 to 1.84] | 1.40 [1.20 to 1.60]
  3-month follow-up: number analyzed (Participants) | 3911 | 3700
  3-month follow-up | 0.16 [0.05 to 0.27] | 0.09 [0.01 to 0.17]
  6-month follow-up: number analyzed (Participants) | 4002 | 3800
  6-month follow-up | 0.69 [0.48 to 0.90] | 0.55 [0.40 to 0.70]
  9-month follow-up: number analyzed (Participants) | 3827 | 3684
  9-month follow-up: number analyzed (Group home) | 206 | 208
  9-month follow-up | 2.27 [2.04 to 2.50] | 2.35 [2.12 to 2.59]
  12-month follow-up: number analyzed (Participants) | 3831 | 3630
  12-month follow-up: number analyzed (Group home) | 206 | 208
  12-month follow-up | 5.67 [5.38 to 5.95] | 5.75 [5.45 to 6.06]
  15-month follow-up: number analyzed (Participants) | 3807 | 3598
  15-month follow-up: number analyzed (Group home) | 206 | 208
  15-month follow-up | 2.22 [1.99 to 2.45] | 2.35 [2.12 to 2.58]
Statistical Analysis 1: Comparison: Generic Best Practices (GBP) vs Tailored Best Practices (TBP); A Poisson GLMM was fit with a main effect for intervention group, linear and quadratic time trends, and interaction effects between intervention and the time trend variables. The model was adjust for stratification factors, baseline infection incidence, agency and included random intercept for group home; Test type: Superiority; p = 0.89, Test of joint null hypothesis from model — A Wald test was used to test against the null hypothesis that intervention main effect and interaction effects between intervention and time trends were simultaneously zero and assess for differences in the mean trend of infections over follow-up; Bonferroni-adjusted p-value is reported to correct for multiplicity for testing outcomes with 6 combinations of outcomes and subpopulations; The point estimates for intervention main effect, intervention by linear time effect, and for intervention by time^2 interaction effect are described in the paper "Tailored vs. General COVID-19 prevention for adults with mental disabilities residing in group homes: a randomized controlled effectiveness-implementation trial" by Bartels S, Levison JH, Trieu HD, et al., published in 2024 in BMC Public Health, doi:10.1186/s12889-024-18835-w

2. Primary Outcome: Best Practices Fidelity
Description: Best Practices Fidelity is measured by the COVID-19 Best Practices Fidelity Measure developed for this project and refined with input from stakeholders on relevant COVID-19-prevention policies (e.g. number of staff and residents participating in recommended screening, masking, hand washing, and vaccination in the group homes). The Fidelity scale was developed by operationally defining 2-4 items to assess each measure, with items scored on a 5- to 6-point continuum with a rating of 5 or 6 indicating full adherence to the fidelity standard and 1 indicating complete lack of adherence. A home's overall, continuous fidelity score was calculated by averaging measure-specific scores by time period. Each active measure was given equal weight. The percentage scores for each of these measures were then averaged together. The overall fidelity score ranged from a low of 20% (1 out of 5 on each item) to a high of 100% (5 out of 5 on each item).
Time Frame: The outcome will be measured at baseline, 3-, 6-, 9-, 12-, and 15-months post-baseline.
Population: Best Practices Fidelity was measured using a voluntary survey completed only by group home Program Directors who consented to participate at each time point. Participant counts are limited to individuals in homes whose Program Directors contributed survey responses during each time period. Participants were assigned to homes based on where they lived or worked during the study period. Since some staff worked in multiple homes across both arms, the samples are not mutually exclusive.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Group home
Arm/Group | Generic Best Practices (GBP) | Tailored Best Practices (TBP)
Number analyzed (Participants) | 4,338 | 4,375
Number analyzed (Group home) | 199 | 207
score on a scale
  Baseline: number analyzed (Participants) | 3161 | 3141
  Baseline: number analyzed (Group home) | 144 | 152
  Baseline | 82.01 [81.46 to 82.57] | 80.27 [79.75 to 80.79]
  3-month follow-up: number analyzed (Participants) | 3234 | 3555
  3-month follow-up: number analyzed (Group home) | 145 | 167
  3-month follow-up | 85.96 [85.47 to 86.45] | 86.11 [85.65 to 86.56]
  6-month follow-up: number analyzed (Participants) | 3279 | 3875
  6-month follow-up: number analyzed (Group home) | 137 | 170
  6-month follow-up | 84.98 [84.42 to 85.54] | 86.14 [85.68 to 86.60]
  9-month follow-up: number analyzed (Participants) | 3232 | 3475
  9-month follow-up: number analyzed (Group home) | 146 | 165
  9-month follow-up | 84.58 [84.07 to 85.09] | 85.24 [84.78 to 85.69]
  12-month follow-up: number analyzed (Participants) | 3134 | 3353
  12-month follow-up: number analyzed (Group home) | 141 | 158
  12-month follow-up | 84.50 [83.94 to 85.06] | 84.69 [84.17 to 85.22]
  15-month follow-up: number analyzed (Participants) | 3088 | 3428
  15-month follow-up: number analyzed (Group home) | 135 | 165
  15-month follow-up | 84.25 [83.66 to 84.84] | 85.28 [84.78 to 85.78]
Statistical Analysis 1: Comparison: Generic Best Practices (GBP) vs Tailored Best Practices (TBP); A GLMM was fit with a main effect for intervention group, linear and quadratic time trends, and interaction effects between intervention and the time trend variables. The model was adjust for stratification factors, baseline fidelity score, agency and included random intercept for group home; Test type: Superiority; p > .99, Wald test — A Wald test was used to test against the null hypothesis that intervention main effect and interaction effects between intervention and time trends were simultaneously zero and assess for differences in the mean trend of scores over follow-up; [statistical method as in outcome 1, analysis 1]; The point estimates for intervention main effect, intervention by linear time effect, and intervention by time^2 interaction effect are described in the paper "Tailored vs. General COVID-19 prevention for adults with mental disabilities residing in group homes: a randomized controlled effectiveness-implementation trial" by Bartels S, Levison JH, Trieu HD, et al., published in 2024 in BMC Public Health, doi:10.1186/s12889-024-18835-w

3. Primary Outcome: Full COVID-19 Vaccination Status Among Residents
Description: This outcome measure reflects the number of group home (GH) residents who were not fully vaccinated at the beginning of the study (by March 31, 2021) but became fully vaccinated during the study period. Individual-level dates of COVID-19 vaccinations were obtained from records maintained by GH organizations. A person was considered to be fully vaccinated when they received the full dosage of initial immunization(s) as recommended by the CDC during the study, either two initial doses of the Pfizer or Moderna vaccine or one dose of the Johnson & Johnson vaccine. Baseline vaccination rates were established from January 1, 2021, to March 31, 2021.
Time Frame: Assessed from April 1 to the date of vaccination (up to June 30, 2022), up to 15 months for each participant.
Population: Residents with SMI or ID/DD who were not fully vaccinated by March 31, 2021.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Best Practices (GBP) | Tailored Best Practices (TBP)
Number analyzed (Participants) | 492 | 407
Participants | 73 | 77
Statistical Analysis 1: Comparison: Generic Best Practices (GBP) vs Tailored Best Practices (TBP); A Cox frailty model was fit to evaluate differences in the hazard of vaccination uptake between arms separately within the combined population of residents with SMI and ID/DD. This model included a main effect for intervention arm and additionally adjusted for stratification factors, GH agency, and GH-level log-normal frailties; Test type: Superiority; p > .99, Regression, Cox — Bonferroni-adjusted p-value is reported to correct for multiplicity for testing outcomes with 6 combinations of outcomes and subpopulations; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.79 to 1.84]

4. Primary Outcome: Full COVID-19 Vaccination Status Among Staff
Description: This outcome measure reflects the number of group home (GH) staff who were not fully vaccinated at the beginning of the study (by March 31, 2021) but became fully vaccinated during the study period. Individual-level dates of COVID-19 vaccinations were obtained from records maintained by GH organizations. A person was considered to be fully vaccinated when they received the full dosage of initial immunization(s) as recommended by the CDC during the study, either two initial doses of the Pfizer or Moderna vaccine or one dose of the Johnson & Johnson vaccine. Baseline vaccination rates were established from January 1, 2021, to March 31, 2021.
Time Frame: Assessed from April 1 to the date of vaccination (up to June 30, 2022), up to 15 months for each participant.
Population: Staff who were not fully vaccinated by March 31, 2021.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Best Practices (GBP) | Tailored Best Practices (TBP)
Number analyzed (Participants) | 836 | 837
Participants | 467 | 471
Statistical Analysis 1: Comparison: Generic Best Practices (GBP) vs Tailored Best Practices (TBP); A Cox frailty model was fit to evaluate differences in the hazard of vaccination uptake between arms separately within the staff population. This model included a main effect for intervention arm and additionally adjusted for stratification factors, GH agency, and GH-level log-normal frailties; Test type: Superiority; p > .99, Regression, Cox — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.86 to 1.15]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline through 15-month follow-up, totaling 1 year and 6 months.
Description: The adverse event data collected for this study includes COVID-19-related events. All deaths and hospitalizations in the data were caused by COVID-19, meaning deaths and hospitalization unrelated to COVID-19 were not included. Furthermore, the adverse events data only include adverse events for group home residents and not for group home staff.
Arm/Group | Generic Best Practices (GBP) | Tailored Best Practices (TBP)
All-Cause Mortality (participants affected / at risk) | 1/2059 | 1/1777
Serious Adverse Events (participants affected / at risk) | 16/2059 | 11/1777
Other Adverse Events (participants affected / at risk) | 0/2059 | 0/1777
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Best Practices (GBP) (N=2059) | Tailored Best Practices (TBP) (N=1777)
Inpatient hospitalization due to COVID-19 infection (Infections and infestations) | 16 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT04726371/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT04726371/SAP_001.pdf